CLINICAL TRIAL: NCT03923959
Title: Evaluation of Tranexamic Acid Prior to Surgery in the Geriatric Hip Fracture Population for the Reduction of Post-Operative Blood Transfusion
Brief Title: Evaluation of TXA Prior to Surgery in the Geriatric Hip Fracture Population
Acronym: TAHFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lancaster General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LancasterGH
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hip Fractures
Keywords: Blood; Transfusion; Hip; Fracture; Surgery; Replacement; Trauma
MeSH Terms: conditions — Hip Fractures; Fractures, Bone; Wounds and Injuries | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: A prospective, double-blinded, randomized study in the geriatric hip fracture population comparing those who receive intravenous tranexamic acid prior to incision to those who receive a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All OR pharmacists are un-blinded to subject randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Active Comparator): 100 cc normal saline with 1g of tranexamic acid in solution
  Interventions: Drug: Tranexamic Acid Injectable Solution
- Placebo (Placebo Comparator): 100 cc normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Solution — 100 cc normal saline mixed with 1g of tranexamic acid in solution
  Other Names: Cyklokapron
  Arms: Intervention
Other: Placebo — 100 cc normal saline
  Arms: Placebo

SUMMARY:
The overall design of the study is a prospective, double-blinded, randomized study in the geriatric hip fracture population comparing those who receive intravenous tranexamic acid prior to incision to those who receive a placebo.

DETAILED DESCRIPTION:
A significant portion of the geriatric hip fracture population have comorbidities including chronic kidney disease, congestive heart failure, ischemic heart disease, stroke, etc. These patients may be anemic prior to the surgery, and are at increased risk for further blood loss as a result of the fracture and surgical operation. However, intra-operative or post-operative blood transfusions also increase the risk of renal and cardiac complications in this population.

Tranexamic acid (TXA) is an anti-fibrinolytic medication that has transformed total joint replacement management regarding blood loss prevention. Geriatric patients requiring emergent hip fracture repair may significantly benefit from routine administration of TXA prior to the procedure to decrease the risk of blood loss. Thus, treatment may further reduce the percentage of patients who experience blood transfusions and complications associated with transfusions.

The investigators will examine if administration of TXA prior to incision in the geriatric hip fracture patient population decreases the risk of intra-operative or post-operative blood transfusions compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Age > or = to 65 years
3. Hip fracture location within the femoral neck, intertrochanteric, and subtrochanteric regions
4. Indication for one of the following surgical interventions: hemiarthroplasty, total hip replacement, sliding plate and screw fixation, or intramedullary fixation

Exclusion Criteria:

1. Indication for closed reduction or percutaneous screw
2. Allergy to TXA
3. Cerebrovascular accident/stroke, active coronary disease/myocardial infarction, or deep vein thrombosis/pulmonary emboli within one (1) month of the fracture
4. Presence of hypercoaguable disorder, including cancer (active disease), elevated blood homocysteine levels, antiphospholipid antibody syndrome and inherited protein deficiencies (antithrombin III, factor V Leiden, protein S & C deficiencies, prothrombin gene mutation)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 283 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Tocks, DO, Principal Investigator — Penn Medicine / Lancaster General Hospital
Locations (1):
- Lancaster General Heatlh / Penn Medicine, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farrow LS, Smith TO, Ashcroft GP, Myint PK. A systematic review of tranexamic acid in hip fracture surgery. Br J Clin Pharmacol. 2016 Dec;82(6):1458-1470. doi: 10.1111/bcp.13079. Epub 2016 Sep 20. PMID 27492116
- [Background] Eubanks JD. Antifibrinolytics in major orthopaedic surgery. J Am Acad Orthop Surg. 2010 Mar;18(3):132-8. PMID 20190103
- [Background] Ponnusamy KE, Kim TJ, Khanuja HS. Perioperative blood transfusions in orthopaedic surgery. J Bone Joint Surg Am. 2014 Nov 5;96(21):1836-44. doi: 10.2106/JBJS.N.00128. PMID 25378512
- [Background] Kagoma YK, Crowther MA, Douketis J, Bhandari M, Eikelboom J, Lim W. Use of antifibrinolytic therapy to reduce transfusion in patients undergoing orthopedic surgery: a systematic review of randomized trials. Thromb Res. 2009 Mar;123(5):687-96. doi: 10.1016/j.thromres.2008.09.015. Epub 2008 Nov 12. PMID 19007970
- [Background] Carson JL, Duff A, Poses RM, Berlin JA, Spence RK, Trout R, Noveck H, Strom BL. Effect of anaemia and cardiovascular disease on surgical mortality and morbidity. Lancet. 1996 Oct 19;348(9034):1055-60. doi: 10.1016/S0140-6736(96)04330-9. PMID 8874456
- [Background] Fillingham YA, Ramkumar DB, Jevsevar DS, Yates AJ, Shores P, Mullen K, Bini SA, Clarke HD, Schemitsch E, Johnson RL, Memtsoudis SG, Sayeed SA, Sah AP, Della Valle CJ. The Efficacy of Tranexamic Acid in Total Hip Arthroplasty: A Network Meta-analysis. J Arthroplasty. 2018 Oct;33(10):3083-3089.e4. doi: 10.1016/j.arth.2018.06.023. Epub 2018 Jun 27. PMID 30007789
- [Background] Fillingham YA, Ramkumar DB, Jevsevar DS, Yates AJ, Shores P, Mullen K, Bini SA, Clarke HD, Schemitsch E, Johnson RL, Memtsoudis SG, Sayeed SA, Sah AP, Della Valle CJ. The Safety of Tranexamic Acid in Total Joint Arthroplasty: A Direct Meta-Analysis. J Arthroplasty. 2018 Oct;33(10):3070-3082.e1. doi: 10.1016/j.arth.2018.03.031. Epub 2018 Mar 22. PMID 29699826
- [Background] Carling MS, Jeppsson A, Eriksson BI, Brisby H. Transfusions and blood loss in total hip and knee arthroplasty: a prospective observational study. J Orthop Surg Res. 2015 Mar 28;10:48. doi: 10.1186/s13018-015-0188-6. PMID 25889413
- [Background] Alshryda S, Mason J, Sarda P, Nargol A, Cooke N, Ahmad H, Tang S, Logishetty R, Vaghela M, McPartlin L, Hungin AP. Topical (intra-articular) tranexamic acid reduces blood loss and transfusion rates following total hip replacement: a randomized controlled trial (TRANX-H). J Bone Joint Surg Am. 2013 Nov 6;95(21):1969-74. doi: 10.2106/JBJS.L.00908. PMID 24196467
- [Background] Alshryda S, Mason J, Vaghela M, Sarda P, Nargol A, Maheswaran S, Tulloch C, Anand S, Logishetty R, Stothart B, Hungin AP. Topical (intra-articular) tranexamic acid reduces blood loss and transfusion rates following total knee replacement: a randomized controlled trial (TRANX-K). J Bone Joint Surg Am. 2013 Nov 6;95(21):1961-8. doi: 10.2106/JBJS.L.00907. PMID 24196466
- [Background] Benoni G, Lethagen S, Nilsson P, Fredin H. Tranexamic acid, given at the end of the operation, does not reduce postoperative blood loss in hip arthroplasty. Acta Orthop Scand. 2000 Jun;71(3):250-4. doi: 10.1080/000164700317411834. PMID 10919295
- [Background] Rajesparan K, Biant LC, Ahmad M, Field RE. The effect of an intravenous bolus of tranexamic acid on blood loss in total hip replacement. J Bone Joint Surg Br. 2009 Jun;91(6):776-83. doi: 10.1302/0301-620X.91B6.22393. PMID 19483232
- [Background] North WT, Mehran N, Davis JJ, Silverton CD, Weir RM, Laker MW. Topical vs Intravenous Tranexamic Acid in Primary Total Hip Arthroplasty: A Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2016 May;31(5):1022-6. doi: 10.1016/j.arth.2015.11.003. Epub 2015 Nov 10. PMID 26703193
- [Background] Kayupov E, Fillingham YA, Okroj K, Plummer DR, Moric M, Gerlinger TL, Della Valle CJ. Oral and Intravenous Tranexamic Acid Are Equivalent at Reducing Blood Loss Following Total Hip Arthroplasty: A Randomized Controlled Trial. J Bone Joint Surg Am. 2017 Mar 1;99(5):373-378. doi: 10.2106/JBJS.16.00188. PMID 28244907
- [Background] Imai N, Dohmae Y, Suda K, Miyasaka D, Ito T, Endo N. Tranexamic acid for reduction of blood loss during total hip arthroplasty. J Arthroplasty. 2012 Dec;27(10):1838-43. doi: 10.1016/j.arth.2012.04.024. Epub 2012 Jun 14. PMID 22704229
- [Background] Fillingham YA, Kayupov E, Plummer DR, Moric M, Gerlinger TL, Della Valle CJ. The James A. Rand Young Investigator's Award: A Randomized Controlled Trial of Oral and Intravenous Tranexamic Acid in Total Knee Arthroplasty: The Same Efficacy at Lower Cost? J Arthroplasty. 2016 Sep;31(9 Suppl):26-30. doi: 10.1016/j.arth.2016.02.081. Epub 2016 Mar 19. PMID 27113948
- [Background] Gomez-Barrena E, Ortega-Andreu M, Padilla-Eguiluz NG, Perez-Chrzanowska H, Figueredo-Zalve R. Topical intra-articular compared with intravenous tranexamic acid to reduce blood loss in primary total knee replacement: a double-blind, randomized, controlled, noninferiority clinical trial. J Bone Joint Surg Am. 2014 Dec 3;96(23):1937-44. doi: 10.2106/JBJS.N.00060. PMID 25471907
- [Background] Levine BR, Haughom BD, Belkin MN, Goldstein ZH. Weighted versus uniform dose of tranexamic acid in patients undergoing primary, elective knee arthroplasty: a prospective randomized controlled trial. J Arthroplasty. 2014 Sep;29(9 Suppl):186-8. doi: 10.1016/j.arth.2014.01.038. Epub 2014 May 27. PMID 24997651
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was enrolled twice for separate hip fractures, so one of the enrollments was removed.
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 146 | 138
Completed | 73 | 68
Not Completed | 73 | 70
Not completed — Death | 16 | 12
Not completed — Lost to Follow-up | 56 | 56
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Participant enrolled twice for separate hip fractures - one enrollment removed. | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participant enrolled twice for separate hip fractures - one enrollment removed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 146 | 137 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 88.2 (11) | 86.0 (8.7) | 87.2 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 106 | 211
  Male | 41 | 31 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 144 | 136 | 280
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 142 | 134 | 276
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 146 | 137 | 283

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Acute Post-operative Transfusion of Packed Red Blood Cells.
Description: Count of participants with acute post-operative transfusion of packed red blood cells along with the corresponding 95% CI.
Time Frame: 3 Months
Population: All participants who underwent treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: 100 cc normal saline with 1g of tranexamic acid in solution
  Tranexamic Acid Injectable Solution: 100 cc normal saline mixed with 1g of tranexamic acid in solution. Includes administration of pre-operative intravenous tranexamic acid and saline for surgical geriatric hip fracture subjects
- Placebo: 100 cc normal saline
  Placebo: 100 cc normal saline
  Includes administration of pre-operative intravenous saline for surgical geriatric hip fracture subjects
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 146 | 137
Participants | 118 | 111
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.966, Regression, Logistic; Odds Ratio (OR) = 1.013, 95% CI 2-sided [0.5597 to 1.834], Standard Error of Mean 0.307; A two-sample proportion test was also completed; the test utilized an α < 0.049 to account for the O'Brien-Fleming adjustment. The p-value for the two-sample proportion test was 0.966

2. Secondary Outcome: Complication Rate
Description: Determine if participants randomized to TXA experienced increased risk of complications compared to placebo. Complications include number of deep vein thrombosis events, pulmonary emboli events, myocardial infarction events, and cerebral vascular events within 12 weeks post hip fracture surgery.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 146 | 137
Participants | 43 | 30
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.183, Chi-squared — a priori threshold for statistical significance was the standard α = 0.05

3. Secondary Outcome: Hospital Readmission
Description: Determine differences between the groups in 30 day readmission rates.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 146 | 137
Participants | 11 | 8
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.729, Chi-squared — a priori threshold for statistical significance was the standard α = 0.05

4. Secondary Outcome: Mortality Rate
Description: Death within 90 days post hip surgery
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 146 | 137
Participants | 15 | 11
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p = 0.655, Chi-squared — a priori threshold for statistical significance was the standard α = 0.05

5. Secondary Outcome: Length of Stay
Description: Length of stay immediately post study intervention/surgery for hip fracture
Time Frame: From date of study intervention/surgery for hip fracture until the date of discharge or date of death from any cause, whichever came first, assessed up to 34 months.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Treatment: Includes administration of pre-operative intravenous tranexamic acid and saline for surgical geriatric hip fracture subjects
- Placebo: Includes administration of pre-operative intravenous saline for surgical geriatric hip fracture subjects
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 146 | 137
days | 5 (4.1) | 4.8 (3.8)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.7832, t-test, 2 sided — a priori threshold for statistical significance was the standard α = 0.05

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 16/146 | 12/137
Serious Adverse Events (participants affected / at risk) | 3/146 | 1/137
Other Adverse Events (participants affected / at risk) | 69/146 | 57/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=146) | Placebo (N=137)
Hyperglycemia (worsening of condition -> death) (Endocrine disorders) | 1 | 0
Acute infarct in R parietal region (pt released on hospice) (Vascular disorders) | 1 | 0
Post-operative respiratory failure with hypercarbia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Death (General disorders) | 0 | 1 — Pt was demonstrating a general decline. Pt started hospice care and expired due to multiple co-morbidities.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=146) | Placebo (N=137)
Moderate (General disorders) | 25 | 19
Mild (General disorders) | 44 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT03923959/Prot_SAP_000.pdf
  • Informed Consent Form (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/59/NCT03923959/ICF_002.pdf